CLINICAL TRIAL: NCT04988373
Title: Evaluation of the Efficiency of Modified Aligner Appliance With NiTi Springs for Treatment of Mild Crowding Cases in Adults.
Brief Title: Evaluation of the Efficiency of Single Aligner Appliance for Treatment of Mild Crowding Cases in Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-06-2021
Record Dates: First submitted 2021-07-23; First posted 2021-08-03 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Crowding of Anterior Mandibular Teeth
Keywords: Mild crowding; Aligner; Orthodontic treatment; Crowded anterior teeth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single aligner appliance (Experimental): Modified aligner appliance with NiTi springs
  Interventions: Device: Modified aligner appliance
- Traditional fixed appliances (Active Comparator): MBT-prescription of metallic brackets.
  Interventions: Device: Traditional fixed appliance

INTERVENTIONS:
Device: Modified aligner appliance — Patients will be treated using a single aligner appliance with NiTi Springs in order to align their crowding teeth.
  Arms: Single aligner appliance
Device: Traditional fixed appliance — Patients will undergo typical orthodontic treatment using an MBT-prescription of metallic brackets.
  Arms: Traditional fixed appliances

SUMMARY:
36 participants who have mild crowding from the Orthodontic Department at University of Damascus Dental School will be randomly assigned into two groups.

1. In the experimental group, patients will be treated using single aligner appliance in order to align their crowding teeth.
2. Control group will undergo typical orthodontic treatment using an MBT-prescription of metallic brackets.

DETAILED DESCRIPTION:
Most adult patients do not prefer traditional fixed appliances for aesthetic reasons, long treatment duration, and relatively difficult oral care. The current study came in order to evaluate the Efficiency of a new single aligner appliance that is both aesthetic and economical.

ELIGIBILITY:
Inclusion Criteria:

1. Adults patients aged between (16 - 28) years.
2. Class I malocclusion with Mild crowding (1 - 4) mm in the anterior region of the mandibular dental arch
3. All lower teeth are existed (except for third molars).
4. No congenitally missing or extracted teeth (except for third molars)
5. Patients have not undergone previous orthodontic treatment.
6. Patient with good oral hygiene (Plaque Index less than 1).
7. With no severe skeletal discrepancy.

Exclusion Criteria:

1. Bimaxillary dentoalveolar severe protrusion.
2. Any systemic diseases affect teeth movement.
3. Bad oral hygiene.
4. Patient lack of commitment toward follow-up appointments.

Ages: 16 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Duration of Alignment | The assessment is based on calculating days from the beginning of treatment till the end of the alignment stage which is expected to happen within 4 to 6 months
  The time required in days will be calculated from the beginning of treatment till the end of the alignment stage.
Change in Little's Index of Irregularity | T0: immediately before the start of orthodontic treatment; T1: after one month; T2: after two months; T3: after three months; T4: after four months; T5: at the end of the alignment stage (which is expected to occur within 4 to 6 months
  The irregularity of the lower incisors is calculated by measuring the amount of deviations of the anatomic contact points between the six anterior teeth in the horizontal direction in mm, since the sum of these measurements represents the value of the index (Little, 1975). When the sum of these deviations is less than 3 mm, this indicates that the teeth are slightly crowded. When the sum is greater than 10 mm, this indicated very severe crowding.
  The ordinary orthodontic treatment aims to keep this Index less than 1 mm at the end of treatment.
Change in Lower Incisors Inclination | immediately before the start of orthodontic treatment; T1: at the end of the alignment stage which is expected to happen within 4 to 6 months
  The angle between the long axis of the lower Incisors and the mandible plane (Go-Me) will be measured using Cephalometric x ray.

CONTACTS AND LOCATIONS:
Overall Officials: Ziad M Alhafi, DDS, Principal Investigator — MSc student at the Orthodontic Department, University of Damascus Dental; Nada Rajeh, DDS,MSc,PhD, Study Chair — Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrer HG. Protecting the integrity of mandibular incisor position through keystoning procedure and spring retainer appliance. J Clin Orthod. 1975 Aug;9(8):486-94. No abstract available. PMID 1072074
- [Background] Qureshi A. The Inman Aligner for anterior tooth alignment. Dent Update. 2008 Oct;35(8):569-71, 574-6. doi: 10.12968/denu.2008.35.8.569. PMID 19055094
- [Background] Little RM. The irregularity index: a quantitative score of mandibular anterior alignment. Am J Orthod. 1975 Nov;68(5):554-63. doi: 10.1016/0002-9416(75)90086-x. PMID 1059332
- [Background] Hennessy J, Al-Awadhi EA. Clear aligners generations and orthodontic tooth movement. J Orthod. 2016 Mar;43(1):68-76. doi: 10.1179/1465313315Y.0000000004. PMID 25939782
- [Background] Hennessy J, Al-Awadhi EA. Clear aligners generations and orthodontic tooth movement. J Orthod. 2016 Jan 8:1-9. doi: 10.1080/14653125.2015.1108725. Online ahead of print. PMID 26743036
- [Derived] Alhafi ZM, Rajeh N. Evaluation of the effectiveness of modified aligner appliance with nickel-titanium springs in treatment of mild crowding of lower incisors: A randomized controlled clinical trial. J World Fed Orthod. 2022 Aug;11(4):107-113. doi: 10.1016/j.ejwf.2022.04.003. Epub 2022 May 24. PMID 35624004